CLINICAL TRIAL: NCT02854800
Title: Smoking Cessation & Opioid Dependence Treatment Integration: Does Timing Matter?
Brief Title: Smoking Cessation & Opioid Dependence Treatment Integration
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: Pfizer (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Melissa Blank, Assistant Professor, West Virginia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WestVirginiaU; NOT-DA-16-013 (Other: National Institute on Drug Abuse)
Record Dates: First submitted 2016-07-22; First posted 2016-08-03 (Estimated); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Smoking Cessation; Opioid Related Disorders
Keywords: varenicline; buprenorphine
MeSH Terms: conditions — Smoking Cessation; Opioid-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: Participants in all 3 study arms were given the same intervention treatment. Arms differed only by the number of days they had been enrolled in an outpatient opioid dependence program.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Weekly Opioid Tx (Experimental): Participants in this group attended an outpatient opioid clinic once per week. As part of the current study, they received 12-week dosing of varenicline per label recommendations: 0.5mg once daily (Days 1-3), 0.5 mg twice daily (Days 4-7), and 1 mg twice daily (Days 8-84). Pill form/blister pack
  Interventions: Drug: varenicline
- Biweekly Opioid Tx (Experimental): Participants in this group attended an outpatient opioid clinic once bi-weekly. As part of the current study, 12-week dosing of varenicline per label recommendations: 0.5mg once daily (Days 1-3), 0.5 mg twice daily (Days 4-7), and 1 mg twice daily (Days 8-84). Pill form/blister pack
  Interventions: Drug: varenicline
- Monthly Opioid Tx (Experimental): Participants in this group attended an outpatient opioid clinic once per month. As part of the current study, 12-week dosing of varenicline per label recommendations: 0.5mg once daily (Days 1-3), 0.5 mg twice daily (Days 4-7), and 1 mg twice daily (Days 8-84). Pill form/blister pack
  Interventions: Drug: varenicline

INTERVENTIONS:
Drug: varenicline — Participants followed the schedule of dosing that is specified on the label: 0.5 mg once daily (Days 1-3), 0.5 mg twice daily (Days 4-7), and 1 mg twice daily (Days 8-84).
  Other Names: Chantix

SUMMARY:
The primary purpose of this study was to examine the feasibility of integrating a smoking cessation intervention for cigarette smokers enrolled in an outpatient program for opioid dependence. The secondary purpose was to compare treatment effects as a function of phase in the outpatient program: 0-90 days (weekly attendance), 90 days-1 year (biweekly attendance), and more than 1 year (monthly attendance).

DETAILED DESCRIPTION:
Tobacco smoking rates are substantially higher among individuals with substance use disorders (SUDs), relative to individuals in the general population (e.g., 97% vs. 19%, respectively). Yet most treatment programs for SUDs fail to address the use of tobacco among patients, and integration of smoking cessation treatment with SUD treatment may improve outcomes for both drugs. The question remains, however, whether to implement a smoking cessation component immediately or only after a patient is stabilized on their SUD pharmacotherapy. Existing research that directly addresses this factor is limited and findings are mixed. Therefore, the purpose of this study was to compare drug use outcomes among patients at three different stages of their SUD treatment: 0-90 days (weekly clinic attendance), 90 days-1 year (biweekly clinic attendance), and more than 1 year (monthly clinic attendance) of consistent abstinence from illicit drugs. Smokers currently in treatment for opioid dependence, at the WVU Comprehensive Opioid Addiction Treatment (COAT) program, were recruited to participate in this 12-week study. Our goal was to complete 20 patients from each of the three COAT treatment groups. During the 12-week intervention period, individuals continued to attend their regular COAT clinic appointments while following a standard varenicline (Chantix®) dosing regimen and responding to questions daily via text messaging (e.g., adherence to varenicline, use of tobacco, tobacco withdrawal side effects, etc.). The primary outcomes are those relevant to feasibility: 1) recruitment, randomization, and retention, 2) adherence to medication regimen, and 3) compliance with responding to text message-based questions. Secondary outcomes include a comparison of the three COAT treatment groups on 1) relapses for all substances, 2) the proportion of smokers abstinent at each assessment (confirmed with expired air carbon monoxide samples), 3) days until successful cigarette quit day, 4) substance withdrawal and medication side effect symptoms, 5) motivation to quit tobacco, and 6) cigarette quit attempts.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in the Comprehensive Opioid Addiction Treatment (COAT) program
* report smoking >10 cigarettes per day for >1 year
* provide an expired air carbon monoxide (CO) reading of >10 parts/million (ppm)
* report interest in making a quit attempt in the next 1-6 months (Contemplation or Preparation stages via the Stage of Change; Prochaska & Diclemente, 1983)
* willing to try varenicline for smoking cessation

Exclusion Criteria:

* current engagement in any form of tobacco cessation (e.g., pharmacotherapy)
* current use of contraindicated medications (e.g., theophylline, warfarin, insulin)
* Stage of Change category as Precontemplation (no plans to quit), Action (actively trying to quit), or Maintenance (have already quit)
* self-reported seizures in the past year
* untreated cardiovascular disease
* self-report breast-feeding
* pregnancy (verified by urinalysis)
* not within 4 weeks of advancing to the next COAT group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa D Blank, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Chestnut Ridge Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Comprehensive Outpatient Addiction Treatment (COAT) program at Chestnut Ridge Hospital on the campus of West Virginia University. Participants were recruited from the COAT clinic between 7/8/2016 and 2/2/2017.
Pre-assignment Details: All participants that were enrolled (after passing the initial screening and not meeting any of the exclusion criteria) were assigned a group.
Groups:
- Weekly Opioid Tx: Participants in this group attended an outpatient opioid clinic once per week. As part of the current study, 12-week dosing of varenicline per label recommendations: 0.5mg once daily (Days 1-3), 0.5 mg twice daily (Days 4-7), and 1 mg twice daily (Days 8-84). Pill form/blister pack
- Bi-weekly Opioid Tx: Participants in this group attended an outpatient opioid clinic once biweekly. As part of the current study, 12-week dosing of varenicline per label recommendations: 0.5mg once daily (Days 1-3), 0.5 mg twice daily (Days 4-7), and 1 mg twice daily (Days 8-84). Pill form/blister pack
Period: Overall Study
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Started | 32 | 28 | 14
Completed | 12 | 15 | 8
Not Completed | 20 | 13 | 6
Not completed — Protocol Violation | 16 | 11 | 3
Not completed — Withdrawal by Subject | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Baseline analysis population is the same as the assignment in Participant Flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx | Total
Number analyzed (Participants) | 32 | 28 | 14 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.38 (6.66) | 32.68 (6.61) | 36.71 (10.36) | 33.67 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 9 | 36
  Male | 16 | 17 | 5 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 30 | 27 | 14 | 71
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 32 | 27 | 14 | 73
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Expired-air Carbon Monoxide [Mean (Standard Deviation); unit: parts per million (ppm)] | 35.72 (17.40) | 33.69 (12.43) | 33.14 (15.20) | 33.92 (16.21)
Cigarettes Smoked per Day [Mean (Standard Deviation); unit: cigarettes per day] | 23.09 (9.19) | 23.15 (8.34) | 27.00 (9.27) | 23.31 (9.49)
Years Smoking [Mean (Standard Deviation); unit: years] | 12.72 (7.48) | 11.23 (6.38) | 14.73 (10.78) | 12.40 (7.89)
Consecutive Days in Opioid Treatment [Mean (Standard Deviation); unit: days] | 45.65 (132.10) | 145.57 (97.82) | 702.38 (502.62) | 193.08 (319.90)
Cigarette Dependence Score [Mean (Standard Deviation); unit: units on a scale] — Fagerstrom Test for Cigarette Dependence scale. Scores ranging from 0-9 with higher scores indicating greater cigarette dependence.
  units on a scale | 6.84 (1.95) | 6.64 (1.91) | 7.43 (1.99) | 6.93 (1.96)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment, Assignment to Treatment, and Retention Rates
Description: For primary feasibility outcomes, recruitment, assignment to treatment, and retention rates were analyzed using descriptive statistics.
Time Frame: up to 12 weeks
Population: All participants that completed informed consent were included to calculate rates of assignment to treatment (N=88). This is different from the number of participants enrolled (N=74) because n=14 participants provided informed consent but were then found to be ineligible for the study based on initial questionnaires.
Measure: Count of Participants; unit: Participants
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Number analyzed (Participants) | 40 | 33 | 15
Participants
  Recruited and Consented | 40 | 33 | 15
  Assigned to Treatment | 32 | 28 | 14
  Completed 4 Weeks | 20 | 19 | 13
  Completed 8 Weeks | 12 | 15 | 9
  Completed 12 Weeks | 12 | 15 | 8

2. Primary Outcome: Percentage of Days on Which Participants Experienced Each Reason for Attrition
Description: Drug withdrawal and medication side effect ratings were assessed as potential reasons for attrition. This assessment was completed by calculating the mean percentage of days, out of the first four weeks, during which effects were reported by participants who completed the entire 12-week protocol versus participants that dropped out. We limited this analysis to the first four weeks.
Time Frame: up to 4 weeks
Population: Participants that completed the entire 12-week study were compared to those that dropped out before completing to determine potential reasons for attrition.
Measure: Mean (Standard Deviation); unit: percentage of study days
Groups:
- Dropouts: Participants that were enrolled and assigned to treatment, but did not complete the entire 12-week study protocol.
- Completers: Participants that were enrolled and completed the entire 12-week protocol.
Arm/Group | Dropouts | Completers
Number analyzed (Participants) | 39 | 35
percentage of study days
  Nausea | 60.3 (38.0) | 43.4 (35.4)
  Headache | 47.2 (38.4) | 39.8 (32.1)
  Sleep Problems | 37.9 (37.3) | 46.6 (40.0)
  Gas/Constipation | 45.9 (40.0) | 48.9 (37.3)
  Abnormal Dreams | 42.0 (33.7) | 53.7 (38.6)
  Depressed Mood | 39.6 (39.6) | 49.0 (38.0)
  Drowsy | 52.8 (36.4) | 50.3 (36.4)
  Craving | 86.5 (23.2) | 78.1 (28.9)
  Irritability | 72.6 (35.1) | 70.4 (29.8)
  Restlessness | 58.7 (40.7) | 56.7 (37.8)
Statistical Analysis 1: Comparison: Dropouts vs Completers; A separate t-test for each row was used to compare dropouts and completers; Test type: Superiority; p < 0.05, t-test, 2 sided

3. Primary Outcome: Number of Study Days With Protocol Non-Adherence
Description: Medication non-adherence rates: The number of study days on which participants a) self-reported not taking the medication (i.e. provided a response of "no") or b) had a missing medication response (i.e. provided no response) via text message.
  Text-messaging non-adherence rates: The number of study days in which participants failed to respond to one or more assessments measured via text message.
Time Frame: up to 12 weeks
Population: Only data for participants that completed the entire 12-week protocol were analyzed. Data were analyzed as a single group/arm as pre-specified in the protocol.
  N=2940 study days (84 days per participant) was the unit of analysis.
Measure: Number; unit: study days
Units Other Than Participants: Study Days
Groups:
- All Participants Aggregated: 12-week dosing of varenicline per label recommendations: 0.5mg once daily (Days 1-3), 0.5 mg twice daily (Days 4-7), and 1 mg twice daily (Days 8-84). Pill form/blister pack
Arm/Group | All Participants Aggregated
Number analyzed (Participants) | 35
Number analyzed (Study Days) | 2940
study days
  Days with missing text data | 1105
  Days of not taking medication | 40
  Days of not reporting medication use | 305

4. Primary Outcome: Medication Acceptability for Completers
Description: Side effect ratings of nausea, headache, sleep problems, gas/constipation, abnormal dreams, depressed mood, and drowsy; scores ranged from 0-10 and higher scores indicate more severe symptoms.
Time Frame: up to 12 weeks
Population: Only analyzed data for participants that completed the entire 12-week protocol.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Number analyzed (Participants) | 12 | 15 | 8
points on a scale
  Nausea | 2.55 (2.08) | 1.46 (0.84) | 3.09 (3.59)
  Headache | 2.21 (1.76) | 1.61 (1.40) | 1.92 (2.66)
  Sleep Disturbances | 3.35 (2.89) | 2.18 (1.67) | 1.07 (1.60)
  Gas/Constipation | 3.41 (2.65) | 2.30 (1.98) | 2.48 (2.47)
  Abnormal Dreams | 3.42 (2.61) | 2.94 (2.16) | 0.82 (1.03)
  Depressed Mood | 2.94 (2.59) | 2.15 (1.59) | 1.10 (0.90)
  Drowsy | 3.40 (2.56) | 2.05 (1.65) | 2.36 (2.79)
Statistical Analysis 1: Comparison: Weekly Opioid Tx vs Bi-weekly Opioid Tx vs Monthly Opioid Tx; One-way ANOVA was used to compare mean medication side effect ratings across the three arms/groups to determine whether one group had more severe symptoms that may have been related to study dropout; Test type: Superiority; p < 0.05, ANOVA; If the overall F test was significant, Tukey's Honestly Significant Difference post-hoc tests were performed

5. Secondary Outcome: Number of Participants With Cigarette Smoking Quit Attempts and Actual Quit
Description: A quit attempt was defined as at least one study day on which 0 cigarettes smoked was reported via text message. Actual quit rates were determined by biochemically verified cigarette abstinence, which was an expired air carbon monoxide reading of < 8 parts per million (ppm).
Time Frame: Up to 12 weeks
Population: Only analyzed data for participants that completed the entire 12-week protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Number analyzed (Participants) | 12 | 15 | 8
Participants
  Quit Attempt Rates | 2 | 2 | 2
  Quit Rates | 0 | 1 | 2

6. Secondary Outcome: Number of Study Days Until First Cigarette Quit Attempt
Description: A quit attempt was defined as at least one day on which participants reported 0 cigarettes smoked via text message. Reports of >0 cigarettes on subsequent days was indicative of relapse.
Time Frame: up to 12 weeks
Population: For this outcome measure, we include only participants that reported at least one study day on which they smoked 0 cigarettes (i.e., made a quit attempt).
Measure: Mean (Standard Deviation); unit: number of study days
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Number analyzed (Participants) | 2 | 2 | 2
number of study days | 35.5 (24.7) | 11.5 (12.0) | 12.5 (3.5)

7. Secondary Outcome: Cigarettes Smoked Per Day
Description: The number of cigarettes smoked per day were reported via text message by participants daily. These numbers were averaged within weeks to give 12 separate average weekly values for cigarettes per day.
Time Frame: up to 12 weeks
Population: Only data for participants that completed the entire 12-week protocol were analyzed.
Measure: Mean (Standard Error); unit: cigarettes per day
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Number analyzed (Participants) | 12 | 15 | 8
cigarettes per day
  Week 1 | 18.21 (2.80) | 15.53 (1.74) | 16.00 (2.00)
  Week 2 | 14.28 (2.30) | 12.02 (1.40) | 11.18 (2.07)
  Week 3 | 11.90 (2.17) | 10.21 (1.66) | 8.04 (2.10)
  Week 4 | 9.34 (1.95) | 9.58 (1.39) | 8.11 (2.37)
  Week 5 | 9.35 (2.17) | 9.52 (1.63) | 7.91 (2.29)
  Week 6 | 9.21 (1.98) | 9.85 (1.66) | 6.68 (2.01)
  Week 7 | 9.40 (2.13) | 9.45 (1.88) | 7.00 (2.30)
  Week 8 | 8.87 (1.99) | 9.87 (1.80) | 7.13 (2.22)
  Week 9 | 7.98 (1.91) | 9.58 (1.85) | 6.55 (2.10)
  Week 10 | 8.34 (2.04) | 9.47 (1.79) | 6.37 (2.21)
  Week 11 | 7.83 (2.03) | 10.90 (2.03) | 6.83 (2.17)
  Week 12 | 7.35 (2.19) | 10.39 (1.83) | 5.23 (1.66)
Statistical Analysis 1: Comparison: Weekly Opioid Tx vs Bi-weekly Opioid Tx vs Monthly Opioid Tx; Mixed ANOVA was used with Study Week (1-12) as the within-subjects, repeated-measures factor and Group as the between-subjects factor. If the overall F test was significant, Tukey's Honestly Significant Difference post-hoc tests were performed; Test type: Superiority; p < 0.05, ANOVA; If the overall F test was significant, Tukey's Honestly Significant Difference post-hoc tests were performed

8. Secondary Outcome: Drug Withdrawal Ratings
Description: Average self-reported ratings for craving, irritability, restless, alert, bored, calm/relaxed, able to focus, nervous, and other; scores ranged from 0-10 and higher scores indicate higher levels of that withdrawal effect
Time Frame: up to 12 weeks
Population: Only analyzed data for participants that completed the entire 12-week protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Number analyzed (Participants) | 12 | 15 | 8
units on a scale
  Craving | 5.03 (1.85) | 4.55 (1.73) | 4.16 (3.19)
  Irritability | 4.37 (1.87) | 3.09 (1.75) | 2.67 (2.27)
  Restless | 3.67 (2.36) | 1.97 (1.49) | 1.87 (2.05)
  Alert | 6.23 (1.76) | 5.26 (2.17) | 7.98 (1.08)
  Bored | 2.98 (1.64) | 1.72 (1.25) | 1.58 (1.74)
  Calm/Relaxed | 5.12 (2.40) | 4.74 (2.29) | 6.75 (2.18)
  Able to Focus | 6.11 (2.20) | 5.48 (2.12) | 8.08 (0.79)
  Nervous | 2.93 (2.81) | 1.96 (1.65) | 1.62 (2.41)
Statistical Analysis 1: Comparison: Weekly Opioid Tx vs Bi-weekly Opioid Tx vs Monthly Opioid Tx; One-way ANOVA was used for each side effect rating with Group as the between-subjects factor. If the overall F test was significant, Tukey's Honestly Significant Difference post-hoc tests were performed; Test type: Superiority; p < 0.05, ANOVA; If the overall F test was significant, Tukey's Honestly Significant Difference post-hoc tests were performed

9. Secondary Outcome: Expired Air Carbon Monoxide
Description: Expired air carbon monoxide levels were measured for participants every 4 weeks at their in-person study visits, resulting in 4 separate measures across the 12-week period.
Time Frame: up to 12 weeks
Population: Only data for participants that completed the entire 12-week protocol were analyzed.
Measure: Mean (Standard Deviation); unit: parts per million (ppm)
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Number analyzed (Participants) | 12 | 15 | 8
parts per million (ppm)
  Baseline | 46.00 (20.75) | 34.27 (11.60) | 34.25 (13.65)
  Week 4 | 34.18 (14.86) | 30.00 (11.58) | 26.13 (18.34)
  Week 8 | 37.45 (19.93) | 28.60 (12.77) | 25.00 (17.67)
  Week 12 | 34.00 (18.42) | 25.27 (9.55) | 24.63 (15.03)
Statistical Analysis 1: Comparison: Weekly Opioid Tx vs Bi-weekly Opioid Tx vs Monthly Opioid Tx; Data were analyzed via mixed ANOVA whereby Study Visit (1-4) was the repeated-measures factor and Group (weekly, biweekly, monthly) was the between-subjects factor. If the overall F test was significant, Tukey's Honestly Significant Difference post-hoc tests were performed; Test type: Superiority; p < 0.05, ANOVA; If the overall F test was significant, Tukey's Honestly Significant Difference post-hoc tests were performed

10. Secondary Outcome: Number of Participants With Relapse for Illicit Drugs (Opioids, Cocaine, THC, Etc)
Description: Relapse was determined by semi-quantitative urine testing (positive vs negative result). Positive results for illicit drugs were assessed separately (opioids, cocaine, THC, benzodiazepines, amphetamines, and atypical antipsychotics).
Time Frame: up to 12 weeks
Population: Only data for participants that completed the entire 12-week protocol were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Number analyzed (Participants) | 12 | 15 | 8
Participants
  THC | 5 | 2 | 0
  Benzodiazapines | 4 | 1 | 1
  Cocaine | 2 | 1 | 0
  Amphetamine | 1 | 0 | 0
  Atypical antipsychotics | 1 | 0 | 0

11. Secondary Outcome: Readiness to Quit Smoking
Description: The Readiness to Quit Ladder was administered to participants at each of their in-person study visits, for a total of 4 data collections. Participants were asked to indicate their readiness to quit smoking on a scale ranging from 0 (I have no interest in quitting smoking) to 10 (I have already quit smoking).
Time Frame: up to 12 weeks
Population: Only data for participants that completed the entire 12-week protocol were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Number analyzed (Participants) | 12 | 15 | 8
units on a scale
  Baseline | 6.17 (0.83) | 5.87 (1.13) | 5.63 (1.69)
  Week 4 | 7.50 (0.80) | 7.20 (0.86) | 7.88 (1.25)
  Week 8 | 7.50 (0.52) | 7.47 (0.74) | 8.38 (0.74)
  Week 12 | 8.33 (1.07) | 7.53 (0.83) | 8.13 (0.64)
Statistical Analysis 1: Comparison: Weekly Opioid Tx vs Bi-weekly Opioid Tx vs Monthly Opioid Tx; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.05, ANOVA; If the overall F test was significant, Tukey's Honestly Significant Difference post-hoc tests were performed

12. Secondary Outcome: Number of Participants That Moved in Stage of Change for Quitting Smoking
Description: Participants indicated one of the following stages of change at each of their four in-person study visits: Precontemplation (no plans to quit smoking), Contemplation (plans to quit smoking in the next 6 months), Preparation (plans to quit smoking in the next 30 days), Action (currently engaging in quitting smoking), or Maintenance (quit smoking more than 6 months ago).
  Data were quantified by determining the number of participants who moved towards quitting (i.e., moved up one or more stages), the number of participants who moved away from quitting (i.e., moved down one or more stages), and and the number of participants who remained in the same stage.
Time Frame: up to 12 weeks
Population: Only data for participants that completed the entire 12-week protocol were included in analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
Number analyzed (Participants) | 12 | 15 | 8
Participants
  Moved away from quitting | 4 | 1 | 0
  Moved toward quitting | 7 | 6 | 4
  Stayed the same | 1 | 8 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the entire course of participant enrollment in the study (approximately 1 year).
Arm/Group | Weekly Opioid Tx | Bi-weekly Opioid Tx | Monthly Opioid Tx
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/28 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/28 | 0/14
Other Adverse Events (participants affected / at risk) | 0/32 | 0/28 | 0/14

LIMITATIONS AND CAVEATS:
Due to the study's pilot nature, the sample size is relatively small and statistical power is relatively low. High rates of participant dropout were observed, possibly due to medication side effects or the burden of daily assessments for 12 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT02854800/Prot_SAP_000.pdf